CLINICAL TRIAL: NCT02188212
Title: A Clinical Evaluation of Hand-veneered, Porcelain-fused NobelProceraTM Crown Shaded Zirconia and NobelProceraTM Full Contour Crown IPS e.Max CAD on Molars
Brief Title: Nobel Procera Crown Shaded Zirconia and NobelProceraTM Full Contour Crown IPS e.Max CAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-158
Record Dates: First submitted 2014-07-03; First posted 2014-07-11 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2014-07

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NobelProcera Crown Shaded Zirconia (Other): NobelProcera Crown Shaded Zirconia molar
  Interventions: Device: NobelProcera Crown Shaded Zirconia

INTERVENTIONS:
Device: NobelProcera Crown Shaded Zirconia

SUMMARY:
Open, controlled, 5-year, prospective, clinical, multi-center study. A total of 143 adult patients will be treated. Female or male, with an age range from 18 (or age of consent) to 70 years, provided they fulfill the inclusion criteria and need two single tooth restorations on contralateral teeth in the same arch. Each patient will receive in minimum one NobelProceraTM Crown Shaded Zirconia and one NobelProceraTM full contour crown IPS e.max CAD in lithium disilicate on the 1st or 2nd molar randomly allocated to the same tooth position contra-laterally in the maxilla or mandible. The patients will be followed for 5 years after receiving their final prosthetic restorations. Possible dropouts and withdrawals, as well as possible adverse events, will be carefully monitored during the entire investigation period.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 (or age of consent) and less than 70 at the time of inclusion.
* The subject is healthy and compliant with good oral hygiene.
* The subject is in need of at least two paired contalateral single-tooth full coverage molar restorations in the maxilla and/or mandible.
* The subject shall have a stable occlusal relationship with a fully restored, fixed opposing dentition.
* Obtained informed consent from the subject.
* No apical disorder or inflammation of abutment teeth, adjacent and opposing teeth.
* Good gingival / periodontal / periapical status of restoring, opposing and adjacent teeth. Healed situation of soft tissue augmentation is allowed.
* The subject is available for the 5-year term of the investigation.

Exclusion Criteria:

* The subject is not able to give her/his informed consent to participate.
* Alcohol or drug abuse as noted in patient records or in patient history.
* Reason to believe that the treatment might have a negative effect on the patient's total situation (psychiatric problems), as noted in patient records or in patient history.
* An existing condition where acceptable retention of the restoration is impossible to attain
* Mobility of the tooth to be restored.
* Pathologic pocket formation of 4 mm or greater around the tooth to be restored.
* Severe bruxism or other destructive habits.
* Amount of attached soft tissue is insufficient (no attached gingiva on the buccal side of the tooth).
* Health conditions, which do not permit the restorative procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To compare the longevity of single cemented ceramic crowns made with shaded zirconia (NobelProceraTM Shaded Zirconia) and NobelProceraTM full contour crowns IPS e.max CAD lithium disilicate on molars. | yearly up to 5 years

SECONDARY OUTCOMES:
Clinical behaviour (CDA Index, soft tissue behavior) of single cemented ceramic crowns made with shaded zirconia (NobelProceraTM Shaded Zirconia) and NobelProceraTM full contour crowns IPS e.max CAD lithium disilicate on molars. | yearly up to 5 years

OTHER OUTCOMES:
survival rate | yearly, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Wolfarth, Prof, Principal Investigator — University of Aachen, Germany
Locations (1):
- Universitätsklinikum Aachen, Aachen, Germany